CLINICAL TRIAL: NCT03082755
Title: Nighttime Agitation and Restless Legs Syndrome in People With Alzheimer's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-09-0152; R01AG051588-02 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Gabapentin

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a pilot, 8-week, double-blind, placebo-controlled randomized clinical trial of GEn versus placebo, in 136 nursing home residents with nighttime agitation, RLS, and moderate to severe Alzheimer's Disease. A placebo arm will allow for a thorough and systematic assessment of the safety of GEn in this specific patient population. A 2-month post-trial follow-up will assess whether RLS treatment is continued by providers and antipsychotics are reduced.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacy, 40 Acres Pharmacy, will maintain records of group assignment. Each participant's assignment will be kept in a separate, unique file uploaded to a UTBox (secure cloud-based file sharing platform) folder created by 40 Acres Pharmacy. Should emergency unmasking be deemed necessary, the Principal Investigator or Co-Investigator will contact the Chief Pharmacist, Forty Acres Pharmacy, who will allow view-only access to the participant's assignment file in UTBox. Participants, their legally authorized representatives and families, participants' physicians, nursing home staff, investigators, and all study personnel will be masked to group assignment. Emergency unmasking of group assignment is expected to be rare. The Data Safety and Monitoring Board will develop guidelines for emergency unmasking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin Enacarbil (GEn) (Experimental): 1 to 2 GEn tablets (300 mg) will be administered by mouth (PO) once a day in the evening (about 5 pm) for 8 weeks then tapered for 1 week. The study drug will be adjusted up to a maximum dosage of 600 mg as tolerated.
  Interventions: Drug: Gabapentin Enacarbil
- Placebo (Placebo Comparator): 1 to 2 Placebo Oral Tablet(s) will be administered once a day in the evening (about 5 pm) for 8 weeks then tapered for 1 week. The placebo drug will be adjusted up to a maximum dosage of 2 tablets as tolerated.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Gabapentin Enacarbil — 1 to 2 GEn tablets (300 milligrams per tablet) will be administered once a day in the evening (about 5pm) for 8 weeks.
  Other Names: Horizant
  Arms: Gabapentin Enacarbil (GEn)
Drug: Placebo Oral Tablet — 1 to 2 Placebo Oral Tablets will be administered once a day in the evening (about 5pm) for 8 weeks.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Nighttime agitation in persons with Alzheimer's disease causes patient suffering, distresses caregivers, and often results in prescriptions for harmful antipsychotics. Effective treatments are lacking because of limited knowledge of the etiology of nighttime agitation. The investigators propose a clinical trial to better elucidate whether a sleep disorder, restless legs syndrome, may be a mechanism for nighttime agitation, and if treatment with gabapentin enacarbil (Horizant®) reduces nighttime agitation, improves sleep, reduces restless legs syndrome behaviors, and reduces antipsychotic medications.

DETAILED DESCRIPTION:
Nighttime agitation and sleep disturbance in persons with dementia (PWD) causes patient suffering, may accelerate cognitive decline, leads to burdened caregivers, and is costly to manage. Pharmacological interventions are primarily antipsychotics and hypnotics. Effectiveness is unconvincing, and these drugs are associated with falls, strokes, and death. There is a lack of tailored, effective, and sustainable treatments for nighttime agitation and sleep disturbance in PWD. The investigators approach to this problem is innovative because, unlike pharmacological interventions in the past, it tailors the intervention to a treatable condition, restless legs syndrome (RLS), which may be causing the nighttime agitation and sleep disturbance. In previous research, the investigators showed that about 24% of PWD have an undiagnosed sleep disorder, RLS; that RLS was associated with nighttime agitation and sleep disturbance in PWD; and the investigators developed and validated an RLS diagnostic and outcome measure suitable for PWD. In order for the investigators' work to significantly impact standards of clinical practice, evidence is needed on whether RLS behaviors cause nighttime agitation, and if treating RLS behaviors reduces or stops nighttime agitation and improves sleep in PWD. The investigators have chosen gabapentin enacarbil (GEn), as the RLS treatment in this research because it is FDA approved for RLS and has a favorable safety profile. The investigators propose an 8-week, double-blind placebo-controlled randomized clinical trial of GEn versus placebo in 156 community-dwelling and long-term care facility residents with nighttime agitation, sleep disturbance, and RLS. The specific aims of this pilot study are to: 1) Determine the effect of GEn, compared to placebo, on nighttime agitation (primary endpoint) in PWD with RLS. The investigators hypothesize that compared to the placebo control group, the treatment group will have fewer nighttime agitation behaviors. 2) Describe the safety profile of GEn compared to placebo in this population. 3) Estimate the effect size of GEn compared to placebo on nighttime sleep and RLS behaviors. The investigators hypothesize that compared to the placebo control group, the treatment group will have better nighttime sleep and fewer RLS behaviors. 4) Explore whether frequency of RLS behaviors is a causal mechanism for nighttime agitation. The investigators hypothesize that frequency of RLS behaviors will mediate the effect of GEn on nighttime agitation behaviors. The results of this study and future definitive trials have the potential to radically shift and drastically improve standards of clinical practice for assessment and treatment of three highly prevalent, often comorbid conditions in PWD: RLS, nighttime agitation, and sleep disturbance. For scientists, the results may provide insight into the mechanism for nighttime agitation and sleep disturbance in PWD and inform future research. For PWD, the findings may result in less nighttime agitation and discomfort from RLS, improved nighttime sleep, and improved sleep may enhance daytime cognitive functioning and quality of life. Application of the findings into the home setting may result in fewer nursing home admissions for PWD and less caregiver burden because the PWD (and their caregivers) can get more sleep.

COVID-19 Modifications - The impact of COVID-19 social distancing on the well-being of community-dwelling older adults with Alzheimer's disease related dementia and their family caregivers who live with them is unknown. They have been confined to their homes. Social and physical activities may be restricted to television and phone calls, and exposure to bright outdoor light is likely infrequent or absent. Exposure to sunlight and both social and physical activity are critical for healthy sleep patterns. For those with the neuropsychiatric symptom of excessive motor activity, such as agitated pacing, being restricted to the home may cause even greater suffering. In addition, family caregivers may be exhausted, stressed, and burdened, even more than usual, because they have not had access to support services such as adult day care, respite, and senior centers. All of the factors associated with social distancing - lack of understanding of what is happening, inadequate or no caregiver support services, isolation, restricted movement, insufficient sunlight, social and physical activity, caregiver exhaustion, and increased caregiver burden - may adversely impact the wellbeing of older adults with Alzheimer's disease related dementia. Further, because older adults with dementing illness are unable to cognitively and verbally express their distress, it is likely that social distancing will increase agitation behaviors, worsen sleep patterns, and increase the need for antipsychotic and sedating medications to manage agitation behaviors and sleep disturbances. We now examine the impact of social distancing on the well-being of older adults with Alzheimer's disease related dementia and their family caregivers who are living together in community settings. A sample of 30 family caregivers will be recruited for qualitative phone interviews to explore the impact of social distancing on the well-being of older adults with Alzheimer's disease related dementia. The specific aims are to: 1) explore the impact of social distancing on nighttime agitation, sleep patterns, and use of antipsychotics and other sedating medications; and 2) ask caregivers for their recommendations on ways to minimize the impact of social distancing on the well-being of older adults with Alzheimer's disease related dementia and their caregivers.

During the time-period where limitations are placed on in-person interactions, researchers will conduct all recruitment, consent, data collection, and intervention activities with participants using remote procedures rather than any procedure that would require in-person interaction. After the university releases restrictions on in-person research activities, researchers may resume in-person activities and/or continue optional telepresence interactions.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=55 years
* Clinical Dementia Rating (CDR) score of 0.5-3, indicating very mild to severe dementia
* Physician diagnosis of dementia of the Alzheimer's type
* Nighttime agitation, defined as Cohen Mansfield Agitation Inventory, Direct Observation total score >=35
* Opinion of the participant's physician that medication for agitation is appropriate
* RLS diagnosis by study advanced practice nurse (APN) or registered nurse (RN) (in consult with the participant's physician, and the investigators), using the Behavioral Indicators Test-Restless Legs
* Medically stable, defined as unchanged medications within 14 days and the absence of fever or other signs and symptoms of acute illness or delirium (e.g. urinary tract infection, pneumonia) that may cause agitation or interfere with the study protocol
* Able to swallow medication
* Ambulatory, with and without assistance
* If currently being treated for RLS, may be included if still having RLS symptoms/signs and confirmed as appropriate for inclusion by medical review

Exclusion Criteria:

* Received >= 50 morphine milligram equivalents per day (MME/d) in the 14 days prior to the randomization decision, because morphine and GEn taken together have a higher incidence of sedation and dizziness than either drug alone
* Currently being treated for RLS with gabapentin or GEn
* Diagnosis of Parkinson's disease (PD) or any other disorder causing tremor because extrapyramidal symptoms may confound RLS diagnosis and actigraphy
* Receiving gabapentin
* Severe psychosis
* Alcohol consumption because combining alcohol and GEn may increase sedation and other adverse events
* Treatment with GEn is contraindicated, such as when a potential participant is receiving multiple antiepileptic drugs, in the opinion of the study APN or RN, participant's physician, or study medical team
* Failure of past treatment with gabapentin or GEn
* Compromised renal function as indicated by creatinine clearance <15 or on hemodialysis
* Current participation in a clinical trial or in any study that may affect study outcomes
* Determined to be at risk for suicide by the study APN, RN, or participant's physician
* Any condition, that in the opinion of the study APN or RN, participant's physician, or study medical team, makes it medically inappropriate for the patient to enroll in the trial
* Persons living independently in the community without a live-in caregiver (family or hired)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Nighttime Agitation - Cohen Mansfield Agitation Inventory (CMAI) - Direct Observation | Change from baseline at 2 and 8 weeks
  The CMAI, modified for direct nighttime observation, will be used to collect objective data on nighttime agitation. Research Assistants (RAs) continuously observe the persons with dementia and record agitation behaviors every 5 minutes. The measure requires that the RAs first note whether the participant is behaviorally awake or asleep. Sleep is defined as a quiet state with eyes closed. Nighttime agitation behaviors are scored during wake. The RA will directly observe the participant when he, or she, is out of bed and record the observations using the CMAI. After the participant has gone to bed, the RA will observe him, or her, via a video camera placed in the bedroom and a small handheld monitor located in a hallway or room adjacent to the bedroom. The monitor will be shielded from view of non-research personnel when on, and turned off between 5-minute observations. The RAs will endeavor to be as sensitive as possible to the privacy of participants.

SECONDARY OUTCOMES:
Nighttime Agitation - Cohen Mansfield Agitation Inventory (CMAI) - Caregiver Version. | Change from baseline at 2 and 8 weeks
  The same primary caregivers, if possible, on the evening and night shifts will each complete the CMAI Caregiver Version at baseline and 8 weeks.
Nighttime Agitation - Modified Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (mADCS-CGIC). | Change from baseline at 2 and 8 weeks
  The mADCS-CGIC measures clinically meaningful change in the patient's condition relative to baseline on a 7-point Likert scale (markedly worse to markedly improved). The scale was modified to assess items specific to agitation, producing global ratings of change in agitation. This scale will be completed by the study Advanced Practice Nurse (APN) based on physical examination and interviews with nursing home caregivers and persons with dementia (if able).
Sleep Disturbance - Direct Observation | Change from baseline at 2 and 8 weeks
  The RA will continuously observe the participant in the evening and night and note every 5 minutes whether the participant is behaviorally awake or asleep. The sleep disturbance outcome will be collected at baseline and 8 weeks. Sleep and wake will be defined as percent of observations asleep or awake on Night 1, 5 pm-10 pm; and Night 2,10 pm-7am. The investigators have chosen to observe on 2 nights at different times to capture any night-to-night and time of night variability in sleep.
Sleep Disturbance - Behavioral Indicators Test - Restless Legs (BIT-RL) | Change from baseline at 2 and 8 weeks
  The BIT-RL consists of two parts: 1) Behavioral Indicators - direct observations for RLS behaviors, such as kicking or rubbing legs (8 items), and 2) Clinical Indicators - medical history or family informant interview (3 items), interviews with caregivers (2 items), and an interview with the resident with dementia (1 item). The research assistants (RAs) will continuously observe each participant for RLS behaviors for 20 minutes on one evening, between 6 pm and the usual bedtime. The study APN will assess for the Restless Legs Syndrome Clinical Indicators by reviewing the medical records, and interviewing family members, evening and night shift nurses, and participants. One item, leg discomfort (yes or no) requires an answer from the participant with dementia. The APN will assess for discomfort in legs in the evening during the interval when the evening nurses report that the participant with dementia is most restless.
Sleep Disturbance - Micro-Mini Motionlogger® Actigraph | Change from baseline at 2 and 8 weeks
  The micro-mini actigraph is wristwatch-sized accelerometer worn on the wrist. In the investigators' previous studies with over 400 nursing home residents with dementia the investigators have "locked" the actigraph on the participant's wrist with a plastic tie that is comfortable to wear, yet difficult to remove. The actigraph is waterproof and can be left on during showers. Nighttime total sleep time is the main actigraphy sleep outcome. The investigators also will measure other sleep disturbance variables, including nighttime wake after sleep onset, sleep efficiency, sleep latency, and awakenings with the actigraph. Daytime will be defined as 7 am-7 pm, and nighttime will be defined as 7 pm- 7 am. Because the investigators have found that sleep varies in persons with dementia and multiple nights are often needed to obtain a more reliable measure, the investigators will measure sleep for 7 days and nights at baseline and 7 days and nights at 8 weeks.

OTHER OUTCOMES:
Fall Risk and Cognition - Global Rating of Fall Risk (GLORF) | Change from baseline at 2 and 8 weeks
  This is a single question measure: "How do you judge the risk that Mr. or Mrs. X will fall within 6 months - high or low?" asked at baseline, week 2, and week 8 of a nurse or aide with personal knowledge of the resident. If possible, the same nurse, aide, or caregiver will complete the GLORF each week.
Mini-Mental State Examination (MMSE) | Change from baseline at 2 and 8 weeks
  The MMSE (range 0-30) is a 30-item cognitive screen measuring orientation, registration, short-term memory, attention/concentration, language and constructional capacity. The MMSE is a widely used screening test of cognition and takes about 10 minutes to administer to the person with dementia.
Physical Mobility Scale (PMS) | Change from baseline at 2 and 8 weeks
  The Physical Mobility Scale (PMS) is an 8-item performance-based scale routinely used to assess mobility of elderly persons living in long-term care facilities.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Richards, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data have been prepared for sharing with other investigators. All collected individual participant data (IPD) can be accessed at https://dataverse.tdl.org/dataset.xhtml?persistentId=doi:10.18738/T8/GDSFSQ after publication of the main study findings
Time Frame: Data will be made available 6 months after publication of the main study findings and will be available in perpetuity.
Access Criteria: IPD will be publicly available via the following url
URL: https://dataverse.tdl.org/dataset.xhtml?persistentId=doi:10.18738/T8/GDSFSQ

REFERENCES:
- [Derived] Richards K, Morrison J, Wang YY, Rangel A, Loera A, Hanlon A, Lozano A, Kovach C, Gooneratne N, Fry L, Allen R. Nighttime Agitation and Restless Legs Syndrome in Persons With Alzheimer's Disease: Study Protocol for a Double-Blind, Placebo-Controlled, Randomized Trial (NightRest). Res Gerontol Nurs. 2020 Nov 1;13(6):280-288. doi: 10.3928/19404921-20200918-01. Epub 2020 Sep 24. PMID 32966585

DOCUMENTS (1):
  • Informed Consent Form (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT03082755/ICF_000.pdf